CLINICAL TRIAL: NCT04006704
Title: A Study to Assess the Acceptability of Scored Film-coated Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Fixed-dose Combination (FDC) Tablets in HIV 1 Infected Pediatric Participants Aged ≥6 to <12 Years, Using Matching Placebo Tablets
Brief Title: Study to Assess the Acceptability of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (D/C/F/TAF) Fixed-Dose Combination (FDC) Tablets in Human Immunodeficiency Virus Type 1 (HIV-1) Infected Pediatric Participants, Using Matching Placebo Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108636; 2019-001384-68 (EudraCT Number); TMC114FD2HTX1006 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: HIV-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D/C/F/TAF (Whole Placebo Tablet then Split Placebo Tablet) (Experimental): Participants will receive scored film-coated 10 milligram (mg) FDC matching placebo tablets (Intake period 1) swallowed whole followed by FDC of scored film-coated D/C/F/TAF 675/150/200/10 mg matching placebo tablets (Intake period 2) swallowed as a split tablet on Day 1. Both the intakes will be separated by at least 15 minutes.
  Interventions: Drug: D/C/F/TAF FDC placebo
- D/C/F/TAF (Split Placebo Tablet then Whole Placebo Tablet) (Experimental): Participants will receive scored film-coated 10 mg FDC matching placebo tablets (Intake period 1) swallowed as a split tablet followed by FDC of scored film-coated D/C/F/TAF 675/150/200/10 mg matching placebo tablets (Intake period 2) swallowed whole on Day 1. Both the intakes will be separated by at least 15 minutes.
  Interventions: Drug: D/C/F/TAF FDC placebo

INTERVENTIONS:
Drug: D/C/F/TAF FDC placebo — Participants will receive matching placebo tablet (whole and split) of D/C/F/TAF 675/150/200/10 mg FDC on Day 1 as intake period 1 and intake period 2.

SUMMARY:
The primary purpose of this study is to assess the ability to swallow the scored film-coated darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) fixed-dose combination (FDC) tablet, irrespective of the mode of intake (whole and split tablet).

DETAILED DESCRIPTION:
This study will be performed in 24 human immunodeficiency virus type 1 (HIV-1) infected pediatric participants. This study is being conducted to obtain data needed to assist in further pediatric development of D/C/F/TAF by assessing the acceptability of the scored film-coated D/C/F/TAF FDC tablet administered as a matching placebo tablet in a pediatric population. At Day 1, each participant will sequentially take 2 placebo tablets and the sequence of placebo tablet, swallowed whole or as split tablet, is assigned by computer generated randomization. After each intake period (within 15 minutes and before the next intake period, as applicable), participants will be asked to fill out an acceptability questionnaires. Every attempt should be made for the participant to complete the questionnaire (marking the correct box to correspond with their impact of taking the placebo tablet). Caregivers may explain the wording/text in the questionnaire to aid in completion. If a participant and his or her caregiver have difficulties in completing the questionnaire, then the study-site personnel may assist. Primarily ability to swallow the scored film-coated D/C/F/TAF FDC tablet, irrespective of the mode of intake will be assessed. Participants safety will be evaluated throughout the study from signing of the Informed Consent Form (ICF)/Assent Form onwards until the last study-related visit.

ELIGIBILITY:
Inclusion Criteria:

* Have a body weight of at least 25 kilogram (kg) and less than (<) 40 kg
* Has documented chronic human immunodeficiency virus type 1 (HIV-1) infection
* Must be on a stable antiretroviral (ARV) regimen for at least 3 months prior to screening
* Has documented plasma HIV-1 ribonucleic acid (RNA) < 400 copies/milliliter (mL) within 6 months prior to screening
* Parent(s) or their legally acceptable representative must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to allow the child to participate in the study. Assent is also required of children capable of understanding the nature of the study (typically 7 years of age and older)

Exclusion Criteria:

* Any active condition (example, active oral infection [candidiasis], significant physical or psychological disease or other findings during screening) that could prevent the participant from swallowing, or limit or confound the protocol-specified assessments and outcomes or for which, in the opinion of the investigator, participation could compromise the safety or well-being of the participant
* Taking any disallowed therapies
* Is a family member of an employee or investigator of the study site with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or is a family member of an employee of Johnson & Johnson
* Have any known allergies to the excipients of the placebo tablet

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who are Able to Swallow the Scored Film-Coated D/C/F/TAF FDC Tablet Irrespective of Mode of Intake | Day 1
  Ability to swallow the scored film-coated tablet irrespective of mode of intake (whole or split tablet) will be assessed.

SECONDARY OUTCOMES:
Acceptability of Intake of the Whole Tablet by the Participant and by the Caregiver | Day 1
  Acceptability of intake of whole tablet will be assessed based on a 3-point questionnaire indicating how hard/easy it is to swallow the tablet, ('hard', 'neither hard or easy','easy') to take this pill.
Acceptability of Intake of the Split Tablet by the Participant and by the Caregiver | Day 1
  Acceptability of intake of split tablet will be assessed based on a 3-point questionnaire indicating how difficult/easy it was to swallow the tablet ('hard', 'neither hard or easy', 'easy') to take the 2 pieces of this pill.
Acceptability of Daily Intake of the Whole Tablet by the Participant | Day 1
  Acceptability of whole tablet describing how it would be if to take this pill once daily for a longer period ('Not Acceptable', 'Acceptable', 'Good to take' to 'Unable to assess this question').
Acceptability of Daily Intake of the Split Tablet by the Participant | Day 1
  Acceptability of Split tablet describing how it would be if to take this pill once daily for a longer period ("Not Acceptable', 'Acceptable', 'Good to take' to 'Unable to assess this question').
Ease of Splitting the Tablet by the Participant's Caregiver | Day 1
  Ease of splitting the tablet by participant's caregiver will be assessed based on a 3- point questionnaire indicating how difficult was it for the participant's caregiver to break the tablet by hand ('hard', 'ok','easy').
Number of Participants with Swallowing Difficulties as Reported by the Observer | Day 1
  Number of Participants with swallowing difficulties as reported by the observer.
Number of Participants with Adverse Events | Up to 22 Days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (8):
- United States (4):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Emory University, Atlanta, Georgia
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Health Science Center, Houston, Texas
- Spain (4):
  - Hosp. Sant Joan de Deu, Esplugues de Llobregat
  - Hosp. Gral. Univ. Gregorio Marañon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Van Hemelryck S, Van Landuyt E, Hufkens V, Vanveggel S. Assessment of swallowability and acceptability of scored darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) fixed-dose combination (FDC) tablets in HIV-1-infected children aged >/=6 to <12 years, using matching placebo tablets: A randomized study. Antivir Ther. 2024 Apr;29(2):13596535241248282. doi: 10.1177/13596535241248282. PMID 38725258
- See also: Link to results on EudraCT registry. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2019-001384-68/results